CLINICAL TRIAL: NCT01872299
Title: Studies Investigating Co-morbidities Aggravating Heart Failure
Acronym: SICA-HF
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University of Hull (Other); Wroclaw Medical University (Other); IRCCS San Raffaele (Other); Hannover Medical School (Other); Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other); Moscow State University of Medicine and Dentistry (Other); Siberian Branch of the Russian Academy of Medical Sciences (Other); Russian Cardiology Research and Production Center (Other); The University Clinic of Pulmonary and Allergic Diseases Golnik (Other); Silesian Centre for Heart Diseases (Other)
Responsible Party: Principal Investigator, Prof. Stefan D Anker, MD, PhD, Charite University, Berlin, Germany
Other Study IDs: FP7/2007-2013, No. 241558; 241558 (Other Grant/Funding Number: European Commission under the 7th Framework Programme)
Record Dates: First submitted 2013-05-17; First posted 2013-06-07 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Heart Failure; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, DNA, biopsies from fat and muscle.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Control: Healthy control subjects
- Heart failure without co-morbidities: Patients with a clinical diagnosis of chronic heart failure without co-morbidities
- Heart failure with co-morbidities: Patients with a clinical diagnosis of chronic heart failure with co-morbidities
- Type 2 diabetes mellitus: Patients with type 2 diabetes mellitus and without heart failure

SUMMARY:
SICA-HF is a prospective, multicentre, multinational, longitudinal, pathophysiological evaluation study, which is being conducted in 11 centres across six countries. SICA-HF receives funding from the European commission's Seventh Framework Programme (FP7/2007-2013) under grant agreement no. 241558 (SICA-HF) and from the Russian Ministry of Science and Education within the file transfer protocol "R&D in priority fields of the S&T complex of Russia 2007-2012" under state contract number 02.527.11.0007. The aim of SICA-HF is to provide detailed characteristics of co-morbidities of heart failure at baseline and over time, particularly with regards to obesity, cachexia, and type 2 diabetes.

DETAILED DESCRIPTION:
SICA-HF, consisting of outstanding European heart failure clinicians and basic researchers, has accomplished to provide a common platform for the two different research teams. All partners of SICA-HF recruited more than 1462 patients with chronic heart failure, 199 patients with type 2 diabetes without heart failure, and 173 healthy control subjects. Thus, during the last year, a cumulative 91.4% of the target value was achieved for patients with chronic heart failure, 66.3% of the target value for diabetic controls, and 115.3% and thus over-achieving for healthy subjects. The data of all participating centers were collected and entered into the central database. As of this writing, 1469 of all chronic heart failure patients' visits, 255 of diabetic controls' visits, and 167 healthy controls' visits have been entered into the online database. In total, 171 patients have been reported to be deceased; the total number of hospitalizations is 2232.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of heart failure;
* Objective evidence of cardiac dysfunctions as evidenced by at least ONE of the following:

  * left ventricular ejection fraction ≤ 40%;
  * left atrial dimension >4.0 cm (or >2.5 cm/m in height)
  * NT-proBNP >400 pg/ml [>47.3 pmol/l] (or BNP >150 pg/ml)
* Current treatment with loop diuretics;
* Age >18 years;
* Willingness to provide informed consent

Exclusion criteria:

* Congenital heart disease;
* Any life-threatening disease other than heart failure;
* Active malignancy of any type, or history of a malignancy within previous 5 years;
* Previous heart transplantation;
* Intra-venous therapy for heart failure given within the previous 72 hours;
* Severe neuro-muscular disease;
* History of unstable angina, myocardial infarction or stroke within 3 months prior to the study;
* Pregnancy;
* Treatment with immunosuppressive therapy, e.g. steroids for rheumatoid arthritis or obstructive lung disease;
* Significant renal dysfunction, defined as serum creatinine >250 μmol/L [>2.8 mg/dL];
* Severe liver disease, defined as any liver function tests >3 times the upper limit of normal;
* Unable to understand and comply with protocol or to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and controls will be recruited from hospitals' outpatients' departments and/or via advertisements; in-patients are permitted if clinically stable.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2010-03; Primary Completion 2015-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Prevalence, incidence, persistence and phenotype of obesity, cachexia and type 2 diabetes in patients with chronic heart failure. | March 31, 2014

SECONDARY OUTCOMES:
Change in exercise capacity and cardiorespiratory reflex control | March 31, 2014
  To describe patterns of exercise capacity and cardiorespiratory reflex control
Change of body composition and its changes over time | March 31, 2014
  To analyse body composition and its changes over time in patients with chronic heart failure and type 2 diabetes, obesity or cachexia
Incidence and prevalence of sleep-disordered breathing and its impact on the clinical severity in patients with chronic heart failure | March 31, 2014
Impact of impaired vascular reactivity on impaired skeletal muscle metabolic and functional capacity, including its underlying mechanisms | March 31, 2014
Changes of metabolic status in patients with heart failure and type 2 diabetes, obesity and cachexia | March 31, 2014
  To describe the interplay and metabolic signalling pathways between adipose tissue, skeletal muscle, the bone marrow and the heart in patients with heart

CONTACTS AND LOCATIONS:
Overall Officials: Stefan D Anker, MD, PhD, Principal Investigator — Charité- University Medicine Berlin, Campus Virchow Klinikum; Stephan von Haehling, MD, PhD, Study Chair — Charité- University Medicine Berlin, Campus Virchow Klinikum; John Cleland, MD, PhD, Study Chair — University of Hull; Piotr Ponikowski, MD, PhD, Study Chair — Wroclaw Medical University; Giuseppe Rosano, MD, PhD, Study Chair — IRCCS San Raffaele; Jens Jordan, MD, PhD, Study Chair — Hannover Medical School; Eugeniy Shlyakhto, MD, PhD, Study Chair — Almazov Federal Center for Heart, Blood & Endocrinology; Vsevolod Tkachuk, MD, PhD, Study Chair — Lomonosov Moscow State University; Rostislav Karpov, MD, PhD, Study Chair — Institute of Cardiology, Siberian Branch, Russian Academy of Medical Sciences; Yelena Parfyonova, MD, PhD, Study Chair — Russian Cardiology Research and Production Complex; Mitja Lainscak, MD, PhD, Study Chair — University Clinic of Respiratory and Allergic diseases Golnik; Piotr Rozentryt, MD, PhD, Study Chair — Silesian Centre for Heart Diseases
Locations (11):
- Germany (2):
  - Hannover Medical School, Hanover, Hannover
  - Charité- University Medicine Berlin, Campus Virchow Klinikum, Berlin, State of Berlin
- IRCCS San Raffaele, Rome, Rom, Italy
- Poland (2):
  - Wroclaw, Medical University, Wroclaw, Wroclaw
  - Silesian Centre for Heart Diseases, Zabrze, Zabrze
- Russia (4):
  - Russian Cardiology Research and Production Complex, Moscow, Moscow
  - Lomonosov Moscow State University, Moscow, Moskow
  - Almazov Federal Center for Heart, Blood & Endocrinology, Saint Petersburg, Sankt-Peterburg
  - Institute of Cardiology, Siberian Branch, Russian Academy of Medical Sciences, Tomsk, Tomsk Oblast
- University Clinic of Respiratory and Allergic diseases Golnik, Golnik, Golnik, Slovenia
- University of HULL, Hull, Hull, United Kingdom

REFERENCES:
- [Background] von Haehling S, Lainscak M, Doehner W, Ponikowski P, Rosano G, Jordan J, Rozentryt P, Rauchhaus M, Karpov R, Tkachuk V, Parfyonova Y, Zaritskey AY, Shlyakhto EV, Cleland JG, Anker SD. Diabetes mellitus, cachexia and obesity in heart failure: rationale and design of the Studies Investigating Co-morbidities Aggravating Heart Failure (SICA-HF). J Cachexia Sarcopenia Muscle. 2010 Dec;1(2):187-194. doi: 10.1007/s13539-010-0013-3. Epub 2010 Dec 17. PMID 21475696
- [Derived] Emami A, Saitoh M, Valentova M, Sandek A, Evertz R, Ebner N, Loncar G, Springer J, Doehner W, Lainscak M, Hasenfuss G, Anker SD, von Haehling S. Comparison of sarcopenia and cachexia in men with chronic heart failure: results from the Studies Investigating Co-morbidities Aggravating Heart Failure (SICA-HF). Eur J Heart Fail. 2018 Nov;20(11):1580-1587. doi: 10.1002/ejhf.1304. Epub 2018 Aug 30. PMID 30160804
- [Derived] Pellicori P, Kallvikbacka-Bennett A, Dierckx R, Zhang J, Putzu P, Cuthbert J, Boyalla V, Shoaib A, Clark AL, Cleland JG. Prognostic significance of ultrasound-assessed jugular vein distensibility in heart failure. Heart. 2015 Jul;101(14):1149-58. doi: 10.1136/heartjnl-2015-307558. Epub 2015 May 25. PMID 26006717
- See also: Study home page — http://www.sica-hf.com/